CLINICAL TRIAL: NCT01989052
Title: A Phase 1/2 Unblinded Trial of Carboxyamidotriazole Orotate (CTO) Alone or in Combination With Lomustine for Bevacizumab-Naïve Adult Patients With Recurrent Malignant Glioma
Brief Title: Ph 1/2 CTO With Lomustine for Bevacizumab-Naive Recurrent Glioma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: This study was terminated early due to funding issues prior to completion of phase I
Sponsor: Annick Desjardins (Other)
Collaborators: Tactical Therapeutics, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Annick Desjardins, Associate Professor of Medicine, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00047969
Record Dates: First submitted 2013-10-21; First posted 2013-11-20 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2016-08

CONDITIONS: Malignant Glioma (WHO Grade III or IV)
Keywords: Carboxyamidotriazole Orotate; CTO; Lomustine; N-(2-chloroethyl)-N'-cyclo-hexyl-N-nitrosourea (CCNU); CeeNU; Malignant Glioma; Pro00047969; Desjardins; Duke; The Preston Robert Tisch Brain Tumor Center
MeSH Terms: conditions — Glioma; Lymphoma, Follicular | interventions — Lomustine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Phase 1: CTO and lomustine (Experimental): The combination of CTO with the standard dosing of 100 mg/m2 of lomustine among patients with recurrent malignant glioma (World Health Organization (WHO) grade III or IV) that have not previously received bevacizumab as treatment for their disease
  Interventions: Drug: CTO; Drug: Lomustine
- Phase 2: CTO alone (Experimental): CTO alone at the MTD established in the Phase 1 portion of this study
  Interventions: Drug: CTO
- Phase 2: CTO and lomustine (Experimental): CTO at the same daily dose of as in the CTO alone arm in combination with 110 mg/m2 oral lomustine every 6 weeks
  Interventions: Drug: CTO; Drug: Lomustine
- Phase 2: Lomustine alone (Experimental): Oral lomustine alone at 110 mg/m2 every 6 weeks
  Interventions: Drug: Lomustine

INTERVENTIONS:
Drug: CTO
  Other Names: Carboxyamidotriazole Orotate
  Arms: Phase 1: CTO and lomustine; Phase 2: CTO alone; Phase 2: CTO and lomustine
Drug: Lomustine
  Other Names: CCNU; CeeNU; Gleostine
  Arms: Phase 1: CTO and lomustine; Phase 2: CTO and lomustine; Phase 2: Lomustine alone

SUMMARY:
This is a Phase 1/2 study of the combination of CTO with lomustine in patients with recurrent malignant glioma to be treated at the Preston Robert Tisch Brain Tumor Center (PRTBTC) at Duke. The Primary Objectives are:

* Phase 1: To determine the maximum tolerated dose (MTD) of CTO when combined with lomustine among patients with recurrent malignant glioma (World Health Organization (WHO) grade III or IV) who have not been previously treated with bevacizumab.
* Phase 2: To assess the efficacy of CTO (either in monotherapy or in combination with lomustine) compared to lomustine alone in patients with recurrent WHO grade IV malignant gliomas that have not been previously treated with bevacizumab based upon 6-month progression free survival (PFS6).

Note: This study was terminated early due to funding issues. At the time of termination, the study was still in Phase 1 and no MTD for the combination of CTO and lomustine had been determined for this population. Phase 2 will not proceed.

DETAILED DESCRIPTION:
In the Phase 1 component of the study, we will conduct a dose-escalation study of the combination of CTO with lomustine among patients with recurrent malignant glioma (WHO grade III or IV). All patients will be bevacizumab-naïve. The dose escalation will be a standard "3+3" design to determine the MTD of CTO in combination with lomustine. The Phase 2 portion of this study will be a randomized screening study comparing CTO alone (Arm A) versus CTO with lomustine (Arm B) versus lomustine alone (Arm C) in patients with recurrent WHO grade IV malignant glioma who are bevacizumab-naïve. Subjects will be randomized with a treatment arm allocation ratio of 2:2:1.

Based on the results of patients who have already taken part in Phase 1 of the study, the Principal Investigator has decided to reduce the dose of lomustine used in combination with CTO in this study by 25% of the FDA-approved dose, due to hematologic side effects (side effects related to lower than expected blood counts). Therefore, the dose of lomustine received in combination with CTO is approximately 75% of the standard recommended dose.

Note: This study was terminated early due to funding issues. At the time of termination, the study was still in Phase 1 and no MTD for the combination of CTO and lomustine had been determined for this population. Phase 2 will not proceed.

ELIGIBILITY:
Inclusion Criteria:

* Phase 1 portion: Patients must have recurrent histologically confirmed diagnosis of WHO grade III or IV malignant glioma with no more than 3 prior progressions
* Phase 2 portion: Patients must have recurrent histologically confirmed diagnosis of WHO grade IV malignant glioma (glioblastoma or gliosarcoma) with no more than 3 prior progressions
* Patients should have received optimal surgical management and radiotherapy prior to study enrollment
* Age ≥ 18 years
* Karnofsky Performance Status (KPS) ≥ 70%
* Bi-dimensionally measurable disease as assessed by magnetic resonance imaging based on RANO criteria
* Absolute Neutrophil Count (ANC) ≥ 1000 cells/µl, Platelets ≥ 100,000 cells/µl (without transfusion within 14 days before enrollment)
* Adequate renal function as indicated by the following: Serum creatinine < 1.25 times upper limit of normal or calculated creatinine clearance ≥ 50 ml/minute and urine dipstick for proteinuria < 2+ unless a 24-hour urine protein <1 g of protein is demonstrated
* Prothrombin time (PT) ≤ 1.5 x upper limit of normal (ULN) and activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN within 14 days prior to first study treatment for patients not receiving anti-coagulation. The use of full-dose oral or parenteral anticoagulants is permitted as long as the PT or aPTT is within therapeutic limits (according to the medical standard of the enrolling institution) and the patient has been on a stable dose of anticoagulants for at least two weeks prior to the first study treatment.
* For patients on corticosteroids, they must be on a stable dose for 7 days prior to anticipated start of study drug, and the dose should not be escalated over entry dose level, if clinically possible.
* Signed informed consent approved by the Institutional Review Board
* No evidence of > grade 1 active central nervous system (CNS) hemorrhage on the baseline MRI or CT scan
* Female patients must not be pregnant or breast-feeding. Female patients of childbearing potential (defined as < 2 years after last menstruation or not surgically sterile) must use a highly effective contraceptive method (allowed methods of birth control, [i.e. with a failure rate of < 1% per year] are implants, injectables, combined oral contraceptives, intra-uterine device [intrauterine device (IUD); only hormonal], sexual abstinence or vasectomized partner) during the trial and for a period of > 6 months following the last administration of trial drug(s). Female patients with an intact uterus (unless amenorrhea for the last 24 months) must have a negative serum pregnancy test within 48 hours prior to first study treatment.
* Fertile male patients must agree to use a highly effective contraceptive method (allowed methods of birth control [i.e. with a failure rate of < 1% per year] include a female partner using implants, injectables, combined oral contraceptives, IUDs [only hormonal], sexual abstinence or prior vasectomy) during the trial and for a period of > 6 months following the last administration of trial drugs.

Exclusion Criteria:

* Pregnancy or breastfeeding
* Treated previously with vascular endothelial growth factor (VEGF) or vascular endothelial growth factor receptor (VEGFR) therapies, including antibodies and tyrosine kinase inhibitors
* Prior disease progression on lomustine
* Taking cytochrome P450 3A4 (CYP3A4) inducers and moderate or strong inhibitors. To note: Corticosteroids are allowed, as long as patients have been on a stable dose for 7 days prior to anticipated start of study drug, and the dose should not be escalated over entry dose level, if clinically possible.
* Co-medication that may interfere with study results; e.g. immuno-suppressive agents other than corticosteroids
* Active infection requiring IV antibiotics 7 days before enrollment
* Prior, unrelated malignancy requiring current active treatment with the exception of cervical carcinoma in situ and adequately treated basal cell or squamous cell carcinoma of the skin
* Less than 12 weeks from radiation therapy, unless progressive disease outside of the radiation field or 2 consecutive scans or histopathologic confirmation
* Treated with immunotherapeutic agents, vaccines, or monoclonal antibody (MAb) therapy within 4 weeks before enrollment, unless the patient has recovered from the expected toxic effects of such therapy
* Treated with alkylating agents within 4 weeks before enrollment or treated within 1 week before enrollment with daily or metronomic chemotherapy, unless the patient has recovered from the expected toxic effects of such therapy
* Prior chemotherapy (non-alkylating agents) within 2 weeks before enrollment, unless the patient has recovered from the expected toxic effects of such therapy
* Current, recent (within 4 weeks of the first infusion of this study), or planned use of an experimental drug, unless the patient has recovered from the expected toxic effects of such therapy

Vascular endothelial growth factor (VEGF) Inhibitor-Specific

Exclusion Criteria are:

* Inadequately controlled hypertension (defined as systolic blood pressure > 150 mmHg and/or diastolic blood pressure > 100 mmHg) within 28 days of first study treatment
* Prior history of hypertensive crisis, hypertensive encephalopathy, reverse posterior leukoencephalopathy syndrome (RPLS)
* Prior history of gastrointestinal perforation or abscess
* Clinically significant (i.e. active) cardiovascular disease, for example cerebrovascular accidents ≤ 6 months prior to study enrollment, myocardial infarction ≤ 6 months prior to study enrollment, unstable angina, New York Heart Association (NYHA) Grade II or greater congestive heart failure (CHF), or serious cardiac arrhythmia uncontrolled by medication or potentially interfering with protocol treatment
* History or evidence upon physical/neurological examination of central nervous system disease (e.g. seizures) unrelated to cancer unless adequately controlled by medication or potentially interfering with protocol treatment
* Significant vascular disease (e.g., aortic aneurysm requiring surgical repair or recent arterial thrombosis) within 6 months prior to start of study treatment
* History of pulmonary hemorrhage/hemoptysis ≥ grade 2 (defined as ≥ 2.5 mL bright red blood per episode) within 1 month of first study treatment
* History or evidence of inherited bleeding diathesis or significant coagulopathy at risk of bleeding (i.e. in the absence of therapeutic anticoagulation)
* Current or recent (within 10 days of study enrollment) use of aspirin (>325 mg/day), clopidogrel (>75 mg/day) or equivalent. Prophylactic or therapeutic low molecular weight heparin (LMWH) is allowed
* Surgical procedure (including open biopsy, surgical resection, wound revision, or any other major surgery involving entry into a body cavity) or significant traumatic injury within 28 days prior to first study treatment, or anticipation of need for major surgical procedure during the course of the study
* Minor surgical procedure, e.g. stereotactic biopsy, within 7 days of first study treatment; placement of a vascular access device, within 2 days of first study treatment
* History of intracranial abscess within 6 months prior to first study treatment
* History of active gastrointestinal bleeding within 6 months prior to first study treatment
* Serious, non-healing wound, active ulcer, or untreated bone fracture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2014-05; Primary Completion 2015-03 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Phase 1: Determine the maximum tolerated dose (MTD) of CTO when combined with lomustine | 1 year
  A standard "3+3" design to determine the MTD of CTO in combination with lomustine. Subjects will be administered CTO orally on a continuous daily dosing schedule, while subjects will receive oral lomustine (110 mg/m2) every 6 weeks. Cohorts of 3-6 subjects will accrue at each dose level of CTO, beginning with 225 mg/m2, until MTD is defined. The MTD is the highest dose level at which ≤ 1 out of 6 experienced a dose limiting toxicity (DLT).
  MTD is defined as the highest dose level at which ≤ 1 out of 6 experienced DLT.
Phase 2: Percentage of subjects who remain alive and progression-free at 6 months | 6 months
  Percentage of participants surviving six months from date of randomization without progression of disease. Progression-free survival (PFS) was defined as the time from date of randomization to the date of the first documented progression according to the Response Assessment in Neuro-Oncology (RANO) criteria, or to death due to any cause.

SECONDARY OUTCOMES:
Phase 2: Percentage of subjects who experience a dose-limiting toxicity (DLT) during any cycle of protocol treatment | 2 years
  All toxicities will be collected using Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. DLTs will be defined as any of the following events that are possibly, probably, or definitely attributable to CTO or lomustine:
  Non-hematologic:
  * Nausea/vomiting of Grade 3 or greater despite maximal antiemetic therapy
  * Diarrhea of Grade 3 or greater despite maximal antidiarrheal therapy
  * Any other Grade 3 or 4 non-hematologic toxicity
  Hematologic:
  * Any Grade 4 neutropenia
  * Grade 3 neutropenia associated with fever of any duration or where significant sepsis results
  * Grade 4 thrombocytopenia
Phase 2: Median Overall Survival (OS) | 2 years
  Time in months from date of randomization to date of death due to any cause. Patients alive as of the last follow-up had OS censored at the last follow-up date. Median OS was estimated using a Kaplan-Meier curve.
Phase 2: 12 month Overall Survival (OS) | 12 months
  Percentage of participants surviving 12 months from date of randomization. OS was defined as time from randomization to the date of death due to any cause.
Phase 2: Percentage of subjects with best overall response (BOR) of complete response (CR) and partial response (PR) | 2 years
  Response is based on Response Assessment in Neuro-Oncology (RANO) criteria as determined by investigator assessment. A confirmation of response was not required. Complete Response was defined as complete disappearance on MRI/CT of all enhancing tumor and mass effect, off all corticosteroids (or receiving only adrenal replacement doses), accompanied by a stable or improving neurologic examination, and maintained for at least 4 weeks. Partial Response was defined as greater than or equal to 50% reduction in tumor size on MRI/CT by bi-dimensional measurement, on a stable or decreasing dose of corticosteroids, accompanied by a stable or improving neurologic examination, and maintained for at least 4 weeks.
Phase 2: Median PFS | 2 years
  Time in months from date of randomization to the date of first progression according to RANO criteria, or to death due to any cause. Patients alive who had not progressed as of the last follow-up will have PFS censored at the last follow-up date. Median PFS was estimated using a Kaplan-Meier curve.

CONTACTS AND LOCATIONS:
Overall Officials: Annick Desjardins, MD, FRCPC, Principal Investigator — Duke University
Locations (1):
- The Preston Robert Tisch Brain Tumor Center at Duke, Durham, North Carolina, United States

REFERENCES:
- See also: The Preston Robert Tisch Brain Tumor Center at Duke — http://www.cancer.duke.edu/btc/